CLINICAL TRIAL: NCT04511715
Title: Efficacy and Safety of Intravitreal Bevacizumab for the Improvement of Severe Non-proliferative Diabetic Retinopathy Without DME: a Randomized Clinical Trial
Brief Title: Intravitreal Bevacizumab for Nonproliferative Diabetic Retinopathy
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zahra Rabbani Khah, Head of ophthalmic research center, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 9800
Record Dates: First submitted 2020-08-11; First posted 2020-08-13 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Non-proliferative Diabetic Retinopathy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravitreal Bevacizumab IVB group (Active Comparator)
  Interventions: Drug: Intravitreal Bevacizumab IVB
- undergo regular follow-up for Diabetic Retinopathy (Sham Comparator)
  Interventions: Other: Follow-up with regular examination for determination of DR progression

INTERVENTIONS:
Drug: Intravitreal Bevacizumab IVB — Intravitreal Bevacizumab IVB group (50 eyes) that receive 6 bimonthly IVBs within a period of 10 months following the enrollment
  Arms: Intravitreal Bevacizumab IVB group
Other: Follow-up with regular examination for determination of DR progression — regular examination for determination of DR progression
  Arms: undergo regular follow-up for Diabetic Retinopathy

SUMMARY:
In this randomized clinical trial, 100 eyes with nonproliferative diabetic retinopathy will be included and divided randomly into 2 groups: Intravitreal Bevacizumab group (50 eyes) that receive 6 bimonthly intravitreal bevacizumab, and control group (50 eyes) that undergo regular follow-up for Diabetic Retinopathy. Diabetic macular edema (DME) will be treated independently in all groups by intravitreal bevacizumab. Primary outcome will be the percentage of patients with progression of 2 or more stages through international diabetic retinopathy staging. The secondary measures will be changes in best corrected visual acuity (BCVA) and central macular thickness (CMT), and number of examinations and injection.

ELIGIBILITY:
Inclusion Criteria:

* Presence of severe NPDR with DRSS score more than 53 with or without diabetic macular edema
* Diagnosis of DM (type 1 or 2) with age more than 18 years' old
* Visual acuity from 20/25 to 20/40 according to Snellen chart examination or more than 69 letters according to ETDRS chart

Exclusion Criteria:

* Presence of proliferative diabetic retinopathy features including vitreous hemorrhage or optic disc or retinal neovascularization
* History of retinal laser photocoagulation
* Tractional retinal detachment involving the macula
* Evidence of neovascularization of angle on examination
* Macular edema due to a cause other than DME
* Any ocular condition which may change visual acuity during the study
* History of intravitreal injection of anti-vascular endothelial growth factor agent in past 3 months
* History of any use of intravitreal corticosteroid
* History of major intra-ocular surgery except cataract surgery in the past 6 months
* History of thromboembolic every in the past 3 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with equal or more than 2 stages of progression in diabetic retinopathy staging | 12 months
  Multiple fundus photographs interpreted by a single vitreoretinal surgeon who is blind to the study groups

SECONDARY OUTCOMES:
Best corrected visual acuity | 12 months
  Best corrected visual acuity based on ETDRS letter scale and logMAR
Central retinal thickness | 12 months
  Central retinal thickness according to macular ocular coherence tomography
Number of visits | 12 months
  Number of visits in each time point